CLINICAL TRIAL: NCT04303923
Title: Reference Diameter and Characteristics of Distal Radial Artery by Ultrasonographic Assessement in Korean Patients
Status: Completed | Type: Observational
Sponsor: Wonju Severance Christian Hospital (Other)
Responsible Party: Principal Investigator, Jun-Won Lee, Associate professor, Wonju Severance Christian Hospital
Other Study IDs: DRAUS
Record Dates: First submitted 2020-03-09; First posted 2020-03-11 (Actual); Last update posted 2020-03-12 (Actual); Status verified 2020-03

CONDITIONS: Radial Artery
Keywords: anatomical snuffbox; distal radial artery; radial artery
MeSH Terms: interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Male group: Male patients who performed transthoracic echocardiography with arterial ultrasonography
  Interventions: Procedure: Ultrasonography
- Female group: Female patients who performed transthoracic echocardiography with arterial ultrasonography
  Interventions: Procedure: Ultrasonography

INTERVENTIONS:
Procedure: Ultrasonography — The diameters of both the radial artery and the distal radial artery were measured by ultrasonography.

SUMMARY:
Radial access is recommended as the standard approach for coronary angiography (CAG) and percutaneous coronary intervention (PCI) based on the evidence in which RA reduced mortality and bleeding events compared with femoral access. Recently, the use of distal radial artery (DRA) is rapidly increasing in accordance with the publication of several studies that have shown easy hemostasis, reduced bleeding complications and low arterial occlusion rate via distal radial approach. However, the diameter of DRA is relatively smaller than radial artery (RA) which can limit the widespread use of this access route. Regarding the size discrepancy, there is a lack of evidence to guide which patients are acceptable or not for CAG and PCI. Therefore, the main purpose of this study was to provide the reference diameter of DRA using ultrasonography in Korean patients. The clinical predictors for small DRA also were evaluated.

DETAILED DESCRIPTION:
Radial access is recommended as the standard approach for coronary angiography (CAG) and percutaneous coronary intervention (PCI) based on the evidence in which RA reduced mortality and bleeding events compared with femoral access. Recently, the use of distal radial artery (DRA) is rapidly increasing in accordance with the publication of several studies that have shown easy hemostasis, reduced bleeding complications and low arterial occlusion rate via distal radial approach. However, the diameter of DRA is relatively smaller than radial artery (RA) which can limit the widespread use of this access route. Regarding the size discrepancy, there is a lack of evidence to guide which patients are acceptable or not for CAG and PCI. Therefore, the main purpose of this study was to provide the reference diameter of DRA using ultrasonography in Korean patients. The clinical predictors for small DRA also were evaluated.

Assessment of arterial diameter by ultasonography Patients were lying on the bed with relaxation in an quiet room. The outer diameters of both DRA and RA were assessed by a perpendicular angle using a linear ultrasound probe (3-4-10.8 MHz) and the average values were recorded. The diameter of RA was measured from 2-3 cm above wrist crease. Anatomical landmark for the measurement of DRA was the bony surface area just distal space from extensor pollicis longus tendon in which the DRA was best palpable then runs down between the first metacarpal and second metacarpal bone (just out of anatomical snuffbox area)

ELIGIBILITY:
Inclusion Criteria:

* Patients planned to perform transthoracic echocardiography with arterial ultrasonography

Exclusion Criteria:

* Age under 20-year
* Poor image quality
* repeated measurement

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients planned to perform transthoracic echocardiography with arterial ultrasonography were consecutively enrolled in a single center.
Sampling Method: Non-Probability Sample
Enrollment: 1162 (Actual)
Dates: Start 2017-07-07 (Actual); Primary Completion 2018-04-13 (Actual); Study Completion 2020-02-29 (Actual)

PRIMARY OUTCOMES:
The diameter of distal radial artery | Through ultrasonographic evaluation (within 1 hour)
  Mean diameter of distal radial artery on both left and right hand

SECONDARY OUTCOMES:
The diameter of radial artery | Through ultrasonographic evaluation (within 1 hour)
  Mean diameter of radial artery on both left and right hand
Arterial diameter index | Through ultrasonographic evaluation (within 1 hour)
  Diameter of measure artery divided by body surface area
Proportion of small distal radial artery | Through ultrasonographic evaluation (within 1 hour)
  Proportion of small distal radial artery (<2.3mm)
Predictor for small distal radial artery | Through ultrasonographic evaluation (within 1 hour)
  Clinical predictor associated with small distal radial artery

CONTACTS AND LOCATIONS:
Overall Officials: Jun-Won Lee, MD, PhD, Principal Investigator — Yonsei University Wonju College of Medicine, Wonju Severance Christian Hospital
Locations (1):
- Wonju Severance Christian Hospital, Wŏnju, Gangwon-do, South Korea